CLINICAL TRIAL: NCT05567575
Title: Culturally Adapted Cognitive Behavior Therapy (CBT) Informed Mobile-Application for First Episode Psychosis (FEP). A Feasibility Randomised Controlled Trial
Brief Title: Cognitive Behavior Therapy (CBT) Informed Mobile-Application for First Episode Psychosis
Acronym: TechCare
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TechCare-001
Record Dates: First submitted 2022-10-01; First posted 2022-10-05 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Psychosis
Keywords: Psychosis; mHealth; Techonology; LMICs
MeSH Terms: conditions — Psychotic Disorders | interventions — Cognitive Behavioral Therapy; Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Researchers doing outcome assessments will be kept masked of the treatment allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TechCare (Experimental): Participants in this arm will receive a mobile app based cognitive behavior therapy informed "TechCare" intervention for a period of 12 weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy,
- Wait-List control group: (Active Comparator): Participants in this arm will be offered the intervention once the intervention arm have completed their 3rd month outcome assessment.
  Interventions: Behavioral: Cognitive Behavioral Therapy,

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy, — TechCare is based on the intelligent real time therapy (iRTT) conceptual model proposed by Kelly et al. iRTT relates to the use of mobile technologies to deliver interventions such as CBT, extending beyond assessment of symptoms. The intervention is based on the treatment manual developed by David G. Kingdon and Douglas Turkington. The intervention is informed by evidence based cognitive models of psychosis, where the participant is able to choose from a list of pre-selected digital self-help strategies that are personalised to each participant. For example, the App may incorporate the participant's favourite music in the form of multimedia or YouTube links, which are prompted during symptom elevation. Other examples may include psychoeducation, goal setting, problem-solving, etc., based on common self-help strategies in CBT for Psychosis (CBTp).
  Other Names: Mobile Health

SUMMARY:
Onset of First Episode Psychosis (FEP) is at a young age and is a critical period influencing the long-term course of the disorder. Failure to identify FEP can lead to serious implications such as disruption of education, reduced long-term employment, huge economic burden, and is associated with significantly higher mortality. The prevalence of psychosis increases rapidly from age 14 onwards with a peak incidence in the late teens and early 20s. The aim of the project is to examine the acceptability and feasibility of a mobile phone application-based intervention 'TechCare-PK', for individuals with psychosis in Pakistan. The main objectives are to determine whether appropriate individuals could be identified and recruited to the study and whether the TechCare App would be an acceptable intervention for individuals with psychosis.

DETAILED DESCRIPTION:
Onset of First Episode Psychosis (FEP) is at a young age and is a critical period influencing the long-term course of the disorder. Failure to identify FEP can lead to serious implications such as disruption of education, reduced long-term employment, huge economic burden, and is associated with significantly higher mortality. The prevalence of psychosis increases rapidly from age 14 onwards with a peak incidence in the late teens and early 20s. The aim of the project is to examine the acceptability and feasibility of a mobile phone application-based intervention 'TechCare-PK', for individuals with psychosis in Pakistan. The main objectives are to determine whether appropriate individuals could be identified and recruited to the study and whether the TechCare App would be an acceptable intervention for individuals with psychosis.

Where there are challenges related to distance, inconvenience, being homebound or reluctance to face-to-face interventions, Mobile Health (mHealth) approaches that leverage mobile devices such as cellular phones and smartphones can be used to support healthcare system. Research has found mobile based interventions as highly acceptable to families and may meet carers' needs in respect of information, guidance, professional and emotional support. These services has been considered as a good and easy mode of exchanging information, providing health related education and advice, management of symptoms, to early recognize the complications, giving reassurance and for providing quality services.

Methods:

Study Design: A multi-center single blind Randomised Controlled Trial (RCT) comparing with Treatment as Usual (TAU) with participants with First Episode Psychosis (FEP) to be recruited from different psychiatric units across four cities in Pakistan i.e., Karachi, Lahore, Hyderabad and Rawalpindi, Pakistan. If required additional centers will be added i.e., Quetta, Multan and Peshawar following proper ethics amendments.

Aim The aim of this study is to design, and test culturally adapted mobile based CBT intervention for patients with FEP.

Objectives:

* Develop and refine an app based intervention (TechCare) based on existing culturally adapted intervention for psychosis, using patient and public involvement. The aim is to improve its potential efficacy, establish acceptability of the refined intervention to potential participants and facilitators and establish mobile app based deliverability of the intervention
* To explore the usefulness of TechCare as an acceptable intervention in reducing symptoms of psychosis.
* Undertake an internal pilot to establish recruitment and attrition rates, compliance with protocol and acceptability of the trial design to participants.

The proposed study will consist of three phases. First phase of study will focus on developing the app based intervention (TechCare) through qualitative work. Second phase will test run the application with 6-8 service users and incorporate suggestions and refinement of intervention and in the third phase we will test it in a randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the study will be:
* Male and Females patients diagnosed with FEP- Schizophrenia or Schizoaffective disorder.
* Over the age of 18 years.
* A score of three or more on any of the positive symptoms on the PANSS
* A Minimum score of one on the Calgary Depression scale (CDS)
* Having smart phone and able to use smart phone functions.
* Able to understand written and spoken Urdu.

Exclusion Criteria:

* Exclusions will be any evidence of organic brain disease, clinically significant concurrent medical illness, learning disability.
* unable to use simple functions of an android phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility measures | From baseline to 3rd month (at the end of intervention)
  Feasibility will be determined by recruitment rates, adherence rate and retention rates. The criterion for success of feasibility is to recruit >50% of eligible participants, adherence rate (number of home assignments completed; > 50%) and retention rate of 70%
Acceptability measure | From baseline to 3rd month (at the end of intervention)
  Acceptability will be determined using participant feedback on the use of app

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale | Changes from baseline to week-12
  The Scale will indicate the Positive and Negative Syndrome for Schizophrenia that has been comprised of 30 items. The 30 items of semi structured questionnaire will measure positive syndromes, like delusions, hallucinations and conceptual disorganization whereas negative syndromes include passive or apathetic social avoidance and blunted affect.
Psychotic Symptom Rating Scales (PSYRATS) | Changes from baseline to week-12
  The dimensions of hallucinations and delusions will be measured by a semi structured interview scale . The dimensions of hallucinations and delusions will be measured by a semi structured interview scale
Calgary Depression Scale (CDS) | Changes from baseline to week-12
  The scale is specially designed to measure the depression for Psychosis, consist of nine items (Addington et al., 1990). CDS will indicate the subjective and qualitative dimensions of depression in Schizophrenia.
The Work and Social Adjustment Scale (WSAS) | Changes from baseline to week-12
  Five items scale that measures the perceived impairment of social life, relationships, home management, work and private leisure having scores between 0 to 8 that means 0 (no impairment) and 8 (very severe impairment) with a total score of 40 (Mundt, Marks, Shear, & Greist, 2002).
EuroQol-5 Dimensions EQ5-D | Changes from baseline to week-12
  An instrument measures the health-related quality of life. Quality of life will be measured in five dimensions, including usual activities, anxiety/depression, pain/discomfort, self-care and mobility (Sobocki et al 2007).
Client Service Receipt Inventory (CSRI): | Changes from baseline to week-12
  We will collect information about the use of other health services (including the informal sector faith healers/Imams) using CSRI.

CONTACTS AND LOCATIONS:
Overall Officials: Omair Husain, MD, Principal Investigator — Centre for Addiciton and Mental Health
Locations (2):
- Pakistan (2):
  - Institute of Psychiatry, Rawalpindi, Punjab Province
  - Civil Hospital, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: Undecided